CLINICAL TRIAL: NCT02978183
Title: A Multi-Center, Double-Masked, Randomized, Phase 2 Evaluation of the Effectiveness of ST266 Ophthalmic Drops Compared to Placebo for the Treatment of Allergic Conjunctivitis Using a Modified Conjunctival Allergen Challenge Model
Brief Title: Evaluation of the Effectiveness of ST266 Ophthalmic Drops Compared to Placebo to Treat Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST266-AC-201
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): 1X ST266 dosed 4 times a day for 8 days
  Interventions: Biological: ST266
- Group 2 (Placebo Comparator): Placebo dosed 4 times a day for 8 days
  Interventions: Drug: Saline (0.9% NaCl)

INTERVENTIONS:
Biological: ST266 — One (1) drop of 1X ST266 ophthalmic eye drops will be administered to each eye 4 times a day for 8 days.
  Arms: Group 1
Drug: Saline (0.9% NaCl) — One (1) drop of saline ophthalmic eye drops will be administered to each eye 4 times a day for 8 days.
  Arms: Group 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of ST266 ophthalmic drops compared to placebo for the treatment of the signs and symptoms of allergic conjunctivitis.

DETAILED DESCRIPTION:
The study is a multi-center, double-masked, randomized, placebo-controlled, modified conjunctival allergen challenge (CAC) model. The primary endpoints of ocular itching and conjunctival redness will be evaluated at the subject's final visit. Subjects who meet inclusion criteria will be randomized to one of two treatment groups (1:1). Randomization will be stratified by average post-CAC itching scores at baseline.

Subjects will be evaluated at baseline and on Days 6, 7 and 8.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age of either gender and any race;
* provide written informed consent and sign the HIPAA form;
* be willing and able to follow all instructions and attend all study visits; have a positive history of ocular allergies and a positive skin test reaction to a seasonal AND perennial allergen as confirmed by an allergic skin test;
* be able and willing to avoid all disallowed medication for the appropriate washout period and during the study;
* be able and willing to discontinue wearing contact lenses for at least 72 hours prior to and during the study trial period;
* (for females capable of becoming pregnant) agree to have urine pregnancy testing performed at screening (must be negative) and at the study exit; must not be lactating; and must agree to use a medically acceptable form of birth control throughout the study duration and for at least 14 days prior to instillation of investigational product). Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
* have a calculated visual acuity of 0.7 logMAR or better in each eye as measured using an ETDRS chart;
* have a positive post-CAC reaction;
* have a positive post-CAC reaction in two out of the first three time points;
* be able to self-administer eye drops satisfactorily or have a caregiver at home routinely available for this purpose.

Exclusion Criteria:

* have known contraindications or sensitivities to the use of the investigational product or any of its components;
* have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters (including but not limited to narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, or pterygium);
* have had ocular surgical intervention within 3 months prior to initiating the study or during the study and/or a history of refractive surgery within the past 6 months;
* have a known history of retinal detachment, diabetic retinopathy, or active retinal disease;
* have the presence of an active ocular infection (bacterial, viral or fungal) or positive history of an ocular herpetic infection at any visit;
* use any of the disallowed medications during the period indicated prior to and during the study;
* have any significant illness (e.g. any autoimmune disease requiring therapy, severe cardiovascular disease [including arrhythmias]) the investigator feels could be expected to interfere with the subject's health or with the study parameters and/or put the subject at any unnecessary risk (includes but is not limited to: poorly controlled hypertension or poorly controlled diabetes, a history of status asthmaticus, organ transplants, a known history of persistent moderate or severe asthma, or a known history of moderate to severe allergic asthmatic reactions to any of the study allergens);
* manifest signs or symptoms of clinically active allergic conjunctivitis in either eye at the screening visit;
* have planned surgery (ocular or systemic) during the trial period or within 30 days after;
* have used an investigational drug or medical device within 30 days of the study or be concurrently enrolled in another investigational product trial;
* be a female who is currently pregnant, planning a pregnancy, or lactating.
* have cancer or have a history of cancer within the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Andover, Massachusetts
  - Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 34 | 36
Completed | 34 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (13.44) | 47 (13.98) | 45.3 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 15 | 14 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 30 | 32 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 10 | 19
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Iris Color [Number; unit: eyes]
  Black | 0 | 0 | 0
  Blue | 10 | 20 | 30
  Brown | 42 | 44 | 86
  Hazel | 8 | 2 | 10
  Green | 8 | 6 | 14
  Other | 0 | 0 | 0
Allergen Disposition [Count of Participants; unit: Participants]
  Dust Mite | 18 | 16 | 34
  Dog Dander | 4 | 5 | 9
  Cockroach | 1 | 4 | 5
  Cat Dander | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Ocular itching evaluated by the subject. Ocular itching was evaluated on a 0-4 scale (with half unit increments allowed). Lower scores indicated less itching.
Time Frame: Day 7 and 8
Population: Pre-Conjunctival Allergen Challenge not evaluated in subject 1-011 on visit 5B
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge: number analyzed (Participants) | 33 | 36
  Day 7, Pre-Conjunctival Allergen Challenge | 0.508 (0.8373) | 0.139 (0.3131)
  Day 7, 5 Minutes Post Conjunctival Allergen Challenge | 2.485 (0.9533) | 2.535 (1.1070)
  Day 7, 7 Minutes Post Conjunctival Allergen Challenge | 2.559 (0.9887) | 2.576 (1.1113)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 2.434 (0.9320) | 2.458 (1.1124)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 2.154 (0.9415) | 2.181 (1.1520)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 1.838 (0.9960) | 1.910 (1.1482)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 1.529 (0.9103) | 1.722 (1.1707)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 1.346 (0.9435) | 1.583 (1.1164)
  Day 8, pre-Conjunctival Allergen Challenge | 0.449 (0.7405) | 0.167 (0.3827)
  Day 8, 5 Minutes Post Conjunctival Allergen Challenge | 2.816 (0.8968) | 2.618 (0.9847)
  Day 8, 7 Minutes Post Conjunctival Allergen Challenge | 2.787 (0.9316) | 2.625 (0.9865)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 2.588 (0.9903) | 2.604 (1.0357)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 2.309 (0.9654) | 2.299 (1.0804)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 2.081 (0.9389) | 1.986 (1.1354)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 1.765 (0.9573) | 1.819 (1.1158)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 1.493 (0.9262) | 1.590 (1.1167)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.0882, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 5 Minutes Post-CAC; Test type: Superiority; p = 0.8032, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 7 Minutes Post-CAC; Test type: Superiority; p = 0.9003, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 10 Minutes Post-CAC; Test type: Superiority; p = 0.9523, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.9071, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.7509, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.2824, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.4017, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.4497, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.1650, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 5 Minutes Post-CAC; Test type: Superiority; p = 0.3494, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 7 Minutes Post-CAC; Test type: Superiority; p = 0.4781, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.9847, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.9731, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 15: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.6984, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 16: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.6265, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 17: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.7848, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 18: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.5789, ANCOVA — Adjustments for multiplicity were not employed

2. Primary Outcome: Conjunctival Redness
Description: Conjunctival redness evaluated by the investigator. Conjunctival redness was evaluated on a 0-4 scale (with half unit increments allowed). Lower scores indicated less redness.
Time Frame: Day 7 and 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge | 1.103 (0.7541) | 1.028 (0.5818)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 2.125 (0.8817) | 1.958 (0.8814)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 1.897 (0.9714) | 1.882 (0.9073)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 1.926 (1.0308) | 1.771 (0.8481)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 1.875 (1.0005) | 1.743 (0.8377)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 1.816 (1.0323) | 1.681 (0.8775)
  Day 8, Pre-Conjunctival Allergen Challenge | 0.912 (0.6682) | 0.819 (0.4766)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 1.963 (0.7909) | 1.917 (0.7319)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 1.963 (0.8075) | 2.111 (0.7870)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 1.882 (0.8101) | 1.951 (0.8036)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 1.735 (0.8549) | 1.785 (0.8241)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 1.596 (0.8791) | 1.625 (0.7476)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.8165, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 Minutes Post-CAC; Test type: Superiority; p = 0.6590, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.7455, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.9212, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.9509, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.7897, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.3183, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.7604, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.7343, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.1530, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.3307, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.3399, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.5137, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.9962, ANCOVA — Adjustments for multiplicity were not employed

3. Secondary Outcome: Ciliary Redness
Description: Ciliary redness evaluated by the investigator. Ciliary redness was evaluated on a 0-4 scale (with half unit increments allowed). A lower score was indicative of less redness.
Time Frame: Day 7 and 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge | 0.912 (0.6243) | 0.750 (0.5445)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 1.838 (0.8368) | 1.799 (0.8341)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 1.691 (0.9925) | 1.729 (0.8353)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 1.713 (0.9417) | 1.625 (0.8420)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 1.654 (0.9150) | 1.583 (0.7488)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 1.603 (0.9869) | 1.493 (0.8608)
  Day 8, pre-Conjunctival Allergen Challenge | 0.581 (0.6053) | 0.521 (0.4487)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 1.691 (0.8189) | 1.743 (0.7058)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 1.699 (0.7804) | 1.931 (0.7310)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 1.625 (0.8556) | 1.792 (0.7688)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 1.463 (0.9027) | 1.569 (0.7806)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 1.346 (0.8528) | 1.458 (0.8007)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.3259, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 Minutes Post-CAC; Test type: Superiority; p = 0.9785, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.5112, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.7771, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.6232, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.8895, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.8974, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.9604, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 minutes Post-CAC; Test type: Superiority; p = 0.5301, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.0386, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.1034, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.0985, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.2342, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.3016, ANCOVA — Adjustments for multiplicity were not employed

4. Secondary Outcome: Episcleral Redness
Description: Episcleral redness evaluated by the investigator. Episcleral redness was evaluated on a 0-4 scale (with half unit increments allowed). A lower score was indicative of less redness.
Time Frame: Day 7 and 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge | 1.029 (0.6622) | 0.910 (0.5579)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 1.868 (0.8217) | 1.819 (0.8401)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 1.757 (0.9283) | 1.778 (0.8468)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 1.787 (0.9656) | 1.701 (0.8036)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 1.721 (0.9939) | 1.618 (0.7500)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 1.669 (1.0275) | 1.583 (0.8345)
  Day 8, pre-Conjunctival Allergen Challenge | 0.507 (0.5822) | 0.424 (0.4544)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 1.735 (0.8210) | 1.708 (0.6827)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 1.706 (0.8404) | 1.896 (0.7055)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 1.647 (0.8144) | 1.701 (0.7508)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 1.412 (0.8680) | 1.583 (0.7488)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 1.353 (0.8575) | 1.347 (0.7495)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.4927, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 minutes Post-CAC; Test type: Superiority; p = 0.8686, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.5772, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.9700, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.7516, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.9532, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.7522, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.6804, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.6267, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.0976, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.4687, ANCOVA
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.0421, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.6085, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.9634, ANCOVA — Adjustments for multiplicity were not employed

5. Secondary Outcome: Chemosis
Description: Chemosis evaluated by the investigator. Chemosis was evaluated on a 0-4 scale (with half unit increments allowed). A lower score was indicative of less chemosis.
Time Frame: Day 7 and 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge | 0.390 (0.3703) | 0.465 (0.3787)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 0.765 (0.4306) | 0.840 (0.4711)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 0.669 (0.5391) | 0.708 (0.4762)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 0.691 (0.5709) | 0.778 (0.4259)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 0.691 (0.6001) | 0.785 (0.5146)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 0.676 (0.6047) | 0.757 (0.4075)
  Day 8, pre-Conjunctival Allergen Challenge | 0.081 (0.2280) | 0.104 (0.1925)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 0.574 (0.6262) | 0.674 (0.4994)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 0.632 (0.7288) | 0.764 (0.4265)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 0.684 (0.7792) | 0.708 (0.4571)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 0.566 (0.7444) | 0.590 (0.5674)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 0.551 (0.8137) | 0.493 (0.6196)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.3322, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 Minutes Pre-CAC; Test type: Superiority; p = 0.8026, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Pre-CAC; Test type: Superiority; p = 0.9981, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.5645, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.5455, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.6980, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.6115, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.4528, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.7551, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.5318, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.9748, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.7706, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.3414, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.4361, ANCOVA — Adjustments for multiplicity were not employed

6. Secondary Outcome: Eyelid Swelling
Description: Eyelid swelling evaluated by the subject. Eyelid swelling was evaluated on a 0-4 scale in which 0.5 unit increments were not allowed. A lower score was indicative of less swelling.
Time Frame: Day 7 and 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge | 0.45 (0.711) | 0.22 (0.404)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 1.22 (0.889) | 1.39 (0.871)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 1.25 (0.915) | 1.33 (0.837)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 1.06 (0.776) | 1.25 (0.841)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 0.96 (0.711) | 1.22 (0.857)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 0.79 (0.780) | 0.97 (0.836)
  Day 8, pre-Conjunctival Allergen Challenge | 0.41 (0.621) | 0.26 (0.500)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 1.35 (0.744) | 1.21 (0.873)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 1.29 (0.740) | 1.19 (0.881)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 1.12 (0.817) | 1.11 (0.887)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 0.94 (0.766) | 1.10 (0.893)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 0.81 (0.728) | 0.89 (0.887)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.0603, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 minutes Post-CAC; Test type: Superiority; p = 0.4857, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.9815, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.6213, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.1831, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.6489, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.2622, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.2397, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.3202, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.2663, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.5672, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.5055, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.8143, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.6901, ANCOVA — Adjustments for multiplicity were not employed

7. Secondary Outcome: Tearing/Watery Eyes
Description: Tearing evaluated by the subject. Tearing was evaluated on a 0-4 scale in which 0.5 unit increments were not allowed. A lower score was indicative of less tearing.
Time Frame: Day 7 and 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge | 0.38 (0.707) | 0.21 (0.437)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 1.15 (0.966) | 1.38 (1.024)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 0.88 (1.038) | 1.22 (1.003)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 0.72 (0.898) | 1.07 (0.965)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 0.71 (0.930) | 0.94 (1.034)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 0.65 (0.875) | 0.85 (0.909)
  Day 8, pre-Conjunctival Allergen Challenge | 0.37 (0.810) | 0.28 (0.553)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 1.07 (1.074) | 1.15 (0.970)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 1.04 (1.090) | 1.13 (0.929)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 0.87 (0.864) | 1.01 (0.906)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 0.76 (0.809) | 1.00 (0.956)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 0.65 (0.803) | 0.88 (0.952)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.4032, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 Minutes Post-CAC; Test type: Superiority; p = 0.2946, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.2863, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.0891, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.5347, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.3733, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.2506, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.8667, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.7640, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.8008, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.4729, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.4742, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.2922, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.3657, ANCOVA — Adjustments for multiplicity were not employed

8. Secondary Outcome: Rhinorrhea
Description: Rhinorrhea evaluated by the subject. Rhinorrhea was evaluated on a 0-4 scale in which 0.5 unit increments were not allowed. A lower score was indicative of less severity.
Time Frame: Day 7 and 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge | 0.33 (0.595) | 0.19 (0.525)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 1.35 (1.152) | 1.47 (1.134)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 1.18 (0.904) | 1.31 (1.142)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 0.97 (0.870) | 0.97 (1.082)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 0.85 (0.821) | 0.89 (1.090)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 0.85 (0.784) | 0.94 (1.068)
  Day 8, pre-Conjunctival Allergen Challenge | 0.29 (0.579) | 0.22 (0.591)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 1.29 (0.938) | 1.39 (1.225)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 1.26 (0.963) | 1.31 (1.283)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 1.09 (0.933) | 1.08 (1.156)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 1.00 (0.853) | 0.92 (1.180)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 0.94 (0.776) | 0.83 (1.108)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.6600, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 minutes Post-CAC; Test type: Superiority; p = 0.6877, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.3340, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.7874, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.3812, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.6987, ANCOVA
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.6832, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.8521, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.7516, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.6252, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.8321, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.8173, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.5445, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.6810, ANCOVA — Adjustments for multiplicity were not employed

9. Secondary Outcome: Nasal Pruritus
Description: Nasal Pruritus evaluated by the subject. Nasal pruritus was evaluated on a 0-4 scale in which 0.5 unit increments were not allowed. A lower score was indicative of less severity.
Time Frame: Day 7 and 8
Population: Pre-Conjunctival Allergen Challenge not evaluated in subject 1-011 on visit 5B
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge: number analyzed (Participants) | 33 | 36
  Day 7, Pre-Conjunctival Allergen Challenge | 0.30 (0.467) | 0.06 (0.232)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 1.03 (1.141) | 1.11 (1.116)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 0.91 (0.965) | 1.03 (1.082)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 0.76 (0.923) | 0.89 (0.950)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 0.76 (0.890) | 0.83 (0.971)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 0.65 (0.774) | 0.75 (0.967)
  Day 8, pre-Conjunctival Allergen Challenge | 0.24 (0.554) | 0.14 (0.487)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 1.03 (1.167) | 0.94 (1.145)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 1.03 (1.087) | 0.83 (1.082)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 0.91 (1.111) | 0.69 (1.009)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 0.68 (0.912) | 0.69 (1.009)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 0.59 (0.821) | 0.64 (1.018)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.0111, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 Minutes Post-CAC; Test type: Superiority; p = 0.3391, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.2390, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.3068, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.4914, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.5185, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.5262, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.6098, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.8849, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.6941, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.5728, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.5931, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.7513, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.7297, ANCOVA — Adjustments for multiplicity were not employed

10. Secondary Outcome: Ear or Palate Pruritus
Description: Ear or palate pruritus evaluated by the subject. Ear or palate pruritus was evaluated on a 0-4 scale in which 0.5 unit increments were not allowed. A lower score was indicative of less severity.
Time Frame: Day 7 and 8
Population: Pre-Conjunctival Allergen Challenge not evaluated in subject 1-011 on visit 5B
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge: number analyzed (Participants) | 33 | 36
  Day 7, Pre-Conjunctival Allergen Challenge | 0.33 (0.595) | 0.19 (0.401)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 1.26 (1.355) | 1.22 (1.245)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 1.18 (1.193) | 1.11 (1.214)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 1.00 (1.073) | 1.08 (1.105)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 0.91 (0.965) | 0.94 (1.094)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 0.88 (0.808) | 0.83 (0.971)
  Day 8, pre-Conjunctival Allergen Challenge | 0.06 (0.239) | 0.19 (0.401)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 1.18 (1.336) | 1.33 (1.352)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 1.15 (1.282) | 1.28 (1.344)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 1.12 (1.274) | 1.19 (1.283)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 1.00 (1.181) | 1.08 (1.204)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 1.00 (1.128) | 0.97 (1.253)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.1259, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 Minutes Post-CAC; Test type: Superiority; p = 0.9234, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.8816, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.5703, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.5428, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.7454, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.8195, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.0909, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.4881, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.3391, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.6065, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.3393, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.8364, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.8858, ANCOVA — Adjustments for multiplicity were not employed

11. Secondary Outcome: Nasal Congestion
Description: Nasal congestion evaluated by the subject. Nasal congestion was evaluated on a 0-4 scale in which 0.5 unit increments were not allowed. A lower score was indicative of less severity.
Time Frame: Day 7 and 8
Population: Pre-Conjunctival Allergen Challenge not evaluated in subject 1-011 on visit 5B
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
score on a scale
  Day 7, Pre-Conjunctival Allergen Challenge: number analyzed (Participants) | 33 | 36
  Day 7, Pre-Conjunctival Allergen Challenge | 0.67 (0.816) | 0.42 (0.906)
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge | 1.44 (1.160) | 1.47 (1.230)
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge | 1.41 (1.048) | 1.36 (1.099)
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge | 1.24 (0.987) | 1.22 (1.072)
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge | 1.15 (0.989) | 1.22 (1.174)
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge | 1.12 (1.008) | 1.17 (1.159)
  Day 8, pre-Conjunctival Allergen Challenge | 0.47 (0.662) | 0.33 (0.717)
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge | 1.29 (1.060) | 1.36 (1.199)
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge | 1.35 (1.070) | 1.39 (1.293)
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge | 1.26 (1.024) | 1.28 (1.279)
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge | 1.18 (0.968) | 1.28 (1.210)
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge | 1.15 (1.048) | 1.22 (1.222)
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: Pre-CAC; Test type: Superiority; p = 0.8818, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 10 minutes Post-CAC; Test type: Superiority; p = 0.8679, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 15 Minutes Post-CAC; Test type: Superiority; p = 0.7856, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 20 Minutes Post-CAC; Test type: Superiority; p = 0.7507, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 25 Minutes Post-CAC; Test type: Superiority; p = 0.8189, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 7: 30 Minutes Post-CAC; Test type: Superiority; p = 0.9206, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 7: All Post-CAC Time Points; Test type: Superiority; p = 0.9591, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: Pre-CAC; Test type: Superiority; p = 0.5302, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 10 Minutes Post-CAC; Test type: Superiority; p = 0.7591, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 15 Minutes Post-CAC; Test type: Superiority; p = 0.8978, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 11: Comparison: Group 1 vs Group 2; Day 8: 20 Minutes Post-CAC; Test type: Superiority; p = 0.7179, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 12: Comparison: Group 1 vs Group 2; Day 8: 25 Minutes Post-CAC; Test type: Superiority; p = 0.7262, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 13: Comparison: Group 1 vs Group 2; Day 8: 30 Minutes Post-CAC; Test type: Superiority; p = 0.8275, ANCOVA — Adjustments for multiplicity were not employed
Statistical Analysis 14: Comparison: Group 1 vs Group 2; Day 8: All Post-CAC Time Points; Test type: Superiority; p = 0.6180, ANCOVA — Adjustments for multiplicity were not employed

12. Secondary Outcome: Nasal Composite Score
Description: A composite score of presence or absence of at least one nasal symptom evaluated by the subject
Time Frame: Day 7 and 8
Population: Pre-Conjunctival Allergen Challenge not evaluated in subject 1-011 on visit 5B
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 34 | 36
Participants
  Day 7, Pre-Conjunctival Allergen Challenge: number analyzed (Participants) | 33 | 36
  Day 7, Pre-Conjunctival Allergen Challenge: Absent | 11 | 23
  Day 7, Pre-Conjunctival Allergen Challenge: PResent | 22 | 13
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge: Absent | 2 | 2
  Day 7, 10 Minutes Post Conjunctival Allergen Challenge: PResent | 32 | 34
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge: Absent | 2 | 2
  Day 7, 15 Minutes Post Conjunctival Allergen Challenge: PResent | 32 | 34
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge: Absent | 3 | 3
  Day 7, 20 Minutes Post Conjunctival Allergen Challenge: PResent | 31 | 33
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge: Absent | 5 | 4
  Day 7, 25 Minutes Post Conjunctival Allergen Challenge: PResent | 29 | 32
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge: Absent | 4 | 4
  Day 7, 30 Minutes Post Conjunctival Allergen Challenge: PResent | 30 | 32
  Day 8, pre-Conjunctival Allergen Challenge: Absent | 18 | 26
  Day 8, pre-Conjunctival Allergen Challenge: PResent | 16 | 10
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge: Absent | 1 | 2
  Day 8, 10 Minutes Post Conjunctival Allergen Challenge: PResent | 33 | 34
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge: Absent | 2 | 3
  Day 8, 15 Minutes Post Conjunctival Allergen Challenge: PResent | 32 | 33
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge: Absent | 4 | 4
  Day 8, 20 Minutes Post Conjunctival Allergen Challenge: PResent | 30 | 32
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge: Absent | 2 | 5
  Day 8, 25 Minutes Post Conjunctival Allergen Challenge: PResent | 32 | 31
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge: Absent | 3 | 6
  Day 8, 30 Minutes Post Conjunctival Allergen Challenge: PResent | 31 | 30
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Day 7: 10 minutes post-CAC; Test type: Superiority; p > 0.9999, Fisher Exact — Adjustments for multiplicity were not employed
Statistical Analysis 2: Comparison: Group 1 vs Group 2; Day 7: 15 minutes post-CAC; Test type: Superiority; p > 0.9999, Fisher Exact — Adjustments for multiplicity will not be employed
Statistical Analysis 3: Comparison: Group 1 vs Group 2; Day 7: 20 minutes post-CAC; Test type: Superiority; p > 0.9999, Fisher Exact — Adjustments for multiplicity will not be employed
Statistical Analysis 4: Comparison: Group 1 vs Group 2; Day 7: 25 minutes post-CAC; Test type: Superiority; p = 0.7312, Fisher Exact — Adjustments for multiplicity will not be employed
Statistical Analysis 5: Comparison: Group 1 vs Group 2; Day 7: 30 minutes post-CAC; Test type: Superiority; p > 0.9999, Fisher Exact — Adjustments for multiplicity will not be employed
Statistical Analysis 6: Comparison: Group 1 vs Group 2; Day 8: 10 minutes post-CAC; Test type: Superiority; p > 0.9999, Fisher Exact — Adjustments for multiplicity will not be employed
Statistical Analysis 7: Comparison: Group 1 vs Group 2; Day 8: 15 minutes post-CAC; Test type: Superiority; p > 0.9999, Fisher Exact — Adjustments for multiplicity will not be employed
Statistical Analysis 8: Comparison: Group 1 vs Group 2; Day 8: 20 minutes post-CAC; Test type: Superiority; p > 0.9999, Fisher Exact — Adjustments for multiplicity will not be employed
Statistical Analysis 9: Comparison: Group 1 vs Group 2; Day 8: 25 minutes post-CAC; Test type: Superiority; p = 0.4297, Fisher Exact — Adjustments for multiplicity will not be employed
Statistical Analysis 10: Comparison: Group 1 vs Group 2; Day 8: 30 minutes post-CAC; Test type: Superiority; p = 0.4791, Fisher Exact — Adjustments for multiplicity will not be employed

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for subjects over a period of 8 days during active treatment. If an AE was unresolved at the final study visit Investigators were instructed to follow-up with subjects until the AE resolved or they were lost to follow-up. If the patient is lost to follow-up, the Investigator should make 3 reasonable attempts to contact the patient via telephone, post, or certified mail.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 2/34 | 3/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=34) | Group 2 (N=36)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 0 (0)
Infected Bite (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT02978183/Prot_002.pdf
  • Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT02978183/SAP_003.pdf